CLINICAL TRIAL: NCT06924632
Title: Phase 3, Multicentre, Randomised, Double-Blinded, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Minoxidil Sublingual (SL) Tablet (2.5 mg) Twice Daily (BID) in the Treatment of Male Androgenetic Alopecia (AGA) in Adults
Brief Title: Efficacy & Safety of Minoxidil SL Tablets in Men With AGA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Samson Clinical Operations Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAM-002
Record Dates: First submitted 2025-04-06; First posted 2025-04-11 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Androgenetic Alopecia; Male Pattern Baldness
Keywords: Hair Loss; Male Pattern Balding
MeSH Terms: conditions — Alopecia | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2.5 mg Sublingual Minoxidil BID (Experimental): 2.5 mg sublingual minoxidil to be taken twice a day, once in the AM and once in the PM.
  Interventions: Drug: Minoxidil
- Placebo BID (Placebo Comparator): placebo to be taken sublingually twice a day, once in the AM and once in the PM.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minoxidil — 2.5 mg Sublingual Minoxidil Tablet
  Arms: 2.5 mg Sublingual Minoxidil BID
Drug: Placebo — Placebo
  Arms: Placebo BID

SUMMARY:
This is a phase 3, multicentre, randomised, double-blinded, placebo-controlled study examining the safety and efficacy of 2.5 mg sublingual (SL) minoxidil tablets taken twice daily in the treatment of androgenetic alopecia (AGA) in men. The duration of study participation is 32 weeks including screening and safety follow up.

The primary efficacy objective is to determine whether treatment with 2.5 mg SL tablets twice daily increases the number of hairs in men with AGA over 24 weeks. The primary safety objective is to evaluate the safety and tolerability of 2.5 mg SL tablets administered twice daily over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender males of at least 18 years of age (inclusive) at the time of Screening.
* In good general health in the opinion of the Investigator.
* Presence of androgenetic alopecia with hair density reduction in the centroparietal area or vertex of the scalp classified as Norwood-Hamilton Type III vertex, IV, V or VI.
* Willing and able to attend all study visits and comply with treatment plan and required study procedures including scalp tattooing and hair trimming.
* Willing to maintain the same hair style, hair colour, and hair length in non-balding areas.
* Able to comprehend and willing to sign and date a written patient informed consent form (PICF).

Exclusion Criteria:

* Norwood-Hamilton Type IIIa, IVa, and Va grades (i.e. participants must have vertex balding).
* Use of topical minoxidil, oral minoxidil, dutasteride, finasteride, drugs with anti-androgenetic or androgenetic properties, or medications that cause hypertrichosis or hypotrichosis within the 6 months prior to enrolment.
* Laser treatment of the scalp within 3 months prior to enrolment.
* History of scalp micropigmentation or hair restoration surgery.
* Use of wigs, hair extensions, hair pieces, or hair weaves at time of enrolment.
* Use of anti-hypertensive medication.
* Current participation in any other investigational drug or medical device trial, which includes administration of an investigational study medication or medical device, or participation in such a trial within 3 months or 5 half-lives of the investigational product, whichever is longer, prior to receiving the first dose.
* History of hypersensitivity or allergies to minoxidil or any of the excipients contained in the study medication.
* Known allergy or sensitivity to tattoo ink.
* Dermatological disorder (e.g. eczema, psoriasis) or infection affecting the target area (vertex or centroparietal area).
* Scalp characteristics, including scarring, that may interfere with examinations.
* Medical condition which adversely affects hair loss.
* Specific underlying conditions (e.g. cardiovascular disease, congestive cardiac failure, cardiac arrhythmia, systemic lupus erythematosus, history of phaeochromocytoma, pulmonary hypertension secondary to mitral stenosis, minoxidil hypersensitivity), clinically significant findings from medical history, clinical laboratory tests, ECG, or vital signs that, in the opinion of the Investigator, could interfere with the objectives of the study or put the participant at risk.
* Moderate to severe renal or hepatic impairment.
* Hypotension (blood pressure less than 90/60 mmHg) or a history of significant symptomatic postural hypotension.
* Untreated or uncontrolled hypertension (blood pressure greater than 150/90 mmHg, not stable on current medication for the past 3 months).
* History or evidence of hair loss other than androgenetic alopecia.
* Unwilling to comply with all study procedures and assessments.
* Scalp hair length less than ~2.5 cm
* History of alcohol and/or substance abuse, or drug-abuse disorders.
* Major surgery within 4 weeks prior to the screening evaluation, or planned surgery prior to completion of all study procedures.
* Site employees or immediate family members of study site employees.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 132 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Non-vellus Target Area Hair Counts (TAHC) | 24 Weeks
  Mean change in the vertex scalp non-vellus TAHC from baseline to week 24.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Premier Specialists Pty Ltd, Kogarah, New South Wales
  - DIRECT, East Melbourne, Victoria
  - DIRECT, Pascoe Vale, Victoria

IPD SHARING:
Plan to Share IPD: No